CLINICAL TRIAL: NCT06181110
Title: Associations Between Actigraphy-Derived Sleep-Wake Patterns and Illness Trajectories and Treatment Response in Major Depressive Disorder
Brief Title: Sleep-Wake Patterns on Illness Trajectories and Treatment Response in MDD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY032
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Depression; Sleep Disorders, Circadian Rhythm
Keywords: Actigraphy; Transdiagnostic Intervention; Depression; Rest-Activity Rhythm
MeSH Terms: conditions — Depression; Sleep Disorders, Circadian Rhythm | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TranS-C Group (Experimental): TranS-C is a personalized, non-pharmacological transdiagnostic intervention that addresses psychosocial, behavioural, and cognitive contributors to sleep and circadian dysfunction. It references the sleep health framework and integrates evidence-based elements, including CBT for insomnia, interpersonal and social rhythm therapy (IPSRT), chronotherapy, and motivation enhancement.
  Interventions: Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction
- Care-As-Usual Group (No Intervention): The participants in this group will not receive the TranS-C treatment but will have access to usual care based on their needs and preferences, including but not limited to pharmacological interventions, psychological interventions, and complementary and alternative medicine. A treatment tracking log will be used to monitor the care the participants receive during the study period. The CAU group will receive self-help TranS-C materials after completing all of the assessments. We will monitor the participants' weekly depression severity using PHQ-9 and refer those who have serious suicidal risk to the PI for further assessment and professional mental health services if deemed necessary.

INTERVENTIONS:
Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction — This intervention is a non-pharmacological approach that targets various factors contributing to sleep and circadian problems. It incorporates evidence-based elements such as CBT for insomnia, IPSRT, chronotherapy, and motivation enhancement. The treatment consists of 8 sessions with 4 cross-cutting modules: case formulation, sleep and circadian education, motivational interviewing, and goal setting. Participants also receive 4 core modules addressing sleep-wake regularity, daytime functioning, correcting beliefs, and maintaining behavioral change. Additionally, 6 optional modules cater to specific sleep-wake patterns, addressing sleep efficiency, excessive time in bed, delayed/advanced sleep phase, sleep-related worry, complex sleep environments, and nightmares. Modules are delivered based on individual needs. Sessions include agenda setting, homework review, treatment content delivery, goal assignment, and session summarization.
  Other Names: TranS-C
  Arms: TranS-C Group

SUMMARY:
The proposed study will include a longitudinal ecological study (Study 1) and a randomised controlled trial (Study 2). The aims will be to (1) identify the sleep-wake profiles in individuals with MDD through clustering; (2) examine the associations between sleep-wake features/profiles and the prognosis of MDD; and (3) investigate the anti-depressant effects of sleep- and circadian-targeted intervention in those with MDD and whether sleep-wake features/profiles may moderate the treatment outcomes. 70 depressed participants from Study 1 will be randomized to Study 2 for the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) group and the care-as-usual (CAU) group in a 1:1 allocation ratio. The study period will be 8 weeks. Major assessments at baseline and immediate post-treatment will be managed by an independent assessor (a research assistant, RA) who is blind to the group allocation. The proposed trial and the nested pilot study will follow the CONSORT and STROBE guidelines, respectively. The intervention will be provided free of charge.The current registration is only for Study 2 of the current research project.

ELIGIBILITY:
Inclusion Criteria for the MDD group:

1. Adults aged 18-65 years living in Hong Kong
2. Being fluent and literate in Cantonese
3. A Patient Health Questionnaire-9 (PHQ-9) score of at least 10, indicating a moderate level of depression.
4. Meeting the DSM diagnostic criteria for current MDD according to the Mini International Neuropsychiatric Interview (MINI)
5. Experiencing ≥ 1 sleep or circadian problem in the past 3 months according to the sleep and circadian problems checklist (i.e., time needed to fall asleep ≥ 30 minutes, wake after sleep onset ≥ 30 minutes, < 6-hour sleep per night or ≥ 9-hour sleep per night per 24-hour period, and falling asleep after 2:00 AM ≥ 3 nights per week; and variability in the sleep-wake schedule ≥ 2.78 hours within a week)
6. Access to an Internet-enabled mobile device (iOS or Android operating system)
7. Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria for the MDD group:

1. Severe medical or neurocognitive disorder(s) that make participation unsuitable based on the team's clinical experience
2. Presence of other psychiatric disorders as assessed by MINI
3. A history of electroconvulsive therapy (ECT)
4. Current involvement in any psychological treatment programme that targets depression and/or sleep and circadian problems
5. A change in the class or dose of any prescribed psychotropic drugs within 6 weeks before the baseline assessment
6. Shift work, pregnancy, or work, family, or other commitments that interfere with regular sleep-wake patterns
7. Presence of other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) based on the cut-off scores of SLEEP-50 (narcolepsy ≥ 7; OSA ≥ 15; RLS/PLMD ≥ 7)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, 8 weekly survey across study 2, and 2 weekly immediate post treatment assessments
  A 9-item questionnaire used for screening, diagnosing, and monitoring the severity of depression.

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, and immediate post treatment assessment
  A 14-item scale measuring anxiety and depression in both hospital and community settings.
Change in Insomnia Severity Index (ISI) | Baseline, and immediate post treatment assessment
  A 7-item scale used to assess the perceived severity of insomnia.
Change in Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) and Sleep-Related Impairment (PROMIS-SRI) | Baseline, 8 weekly survey across study 2, and 2 weekly immediate post treatment assessments
  8-item scales to assess sleep and circadian functions.
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, and immediate post treatment assessment
  A 20-item scale used to assess five dimensions of fatigue.
Change in Short Form (6-Dimension) Health Survey (SF-6D) | Baseline, and immediate post treatment assessment
  A health survey used for measuring the quality of life on six dimensions.
Change in Sheehan Disability Scale (SDS) | Baseline, and immediate post treatment assessment
  A 5-item scale used to assess functional impairments in work/ school, social life, and family life.
Change in Core Consensus Standardized Sleep Diary | 10-week daily survey
  A 9-item scale used to record sleep time, wake time, perceived sleeping quality, and use of hypnotics.

OTHER OUTCOMES:
Change in Treatment Acceptability/ Adherence Scale (TAAS) | Baseline, and immediate post treatment assessment
  A 10-item scale of the willingness to utilize or recommend the intervention.
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, and immediate post treatment assessment
  A 6-item scale used to rate the treatment's credibility, satisfaction, and expectation for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong